CLINICAL TRIAL: NCT00253734
Title: Immunogenicity and Safety of a Split, Inactivated, Trivalent Influenza Vaccine Administered by Intradermal Route Compared to an Intramuscular Vaccination With Fluzone® in Healthy Adults
Brief Title: Immunogenicity and Safety of Different Doses of Fluzone® Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-0109
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2008-07

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (7):
- 4 (Active Comparator): 31 subjects to receive 15 mcg of TIV administered intramuscularly.
  Interventions: Biological: Fluzone® (IM)
- 2 (Experimental): 31 subjects to receive 6 mcg of TIV administered intradermally.
  Interventions: Biological: Fluzone®
- 1 (Experimental): 31 subjects to receive 9 mcg of TIV administered intradermally.
  Interventions: Biological: Fluzone®
- 3 (Experimental): 31 subjects to receive 3 mcg of TIV administered intradermally.
  Interventions: Biological: Fluzone®
- 5 (Active Comparator): 31 subjects to receive 9 mcg of TIV administered intramuscularly.
  Interventions: Biological: Fluzone® (IM)
- 7 (Active Comparator): 31 subjects to receive 3 mcg of TIV administered intramuscularly.
  Interventions: Biological: Fluzone® (IM)
- 6 (Active Comparator): 31 subjects to receive 6 mcg of TIV administered intramuscularly.
  Interventions: Biological: Fluzone® (IM)

INTERVENTIONS:
Biological: Fluzone® (IM) — 15, 9, 6, or 3 mcg of standard trivalent inactivated influenza vaccine (TIV) administered by the standard intramuscular route.
  Arms: 4; 5; 6; 7
Biological: Fluzone® — 9, 6, or 3 mcg of standard trivalent inactivated influenza vaccine (TIV) administered by intradermal route (Mantoux technique).
  Arms: 1; 2; 3

SUMMARY:
The purpose of this research study is to find out if giving the smaller dose of flu vaccine under the skin generates antibodies against flu compared to giving the vaccine the usual way, as a shot in the arm. If using smaller doses in this manner is effective, the current supply of vaccine could be used to make more doses to give to more people. About 217 healthy adults, 18 to 49 years of age, will participate. The study will be conducted at one site in the United States and subjects are expected to participate for about 6 months. Blood samples will be taken to assess the immune system response. Local and systemic safety will be evaluated in the 28 days following vaccination.

DETAILED DESCRIPTION:
This study is a randomized, prospective, active-controlled, single-center, open label, dose-ranging clinical trial of TIV (Fluzone®) administered to healthy 18-to-49 year old adults who did not receive 2003-2004, 2004-2005 and 2005-2006 influenza vaccine. Subjects will be randomized to one of 7 groups (4 intramuscular and 3 intradermal) to compare the immunogenicity and safety of different concentrations of the standard Fluzone® administered intradermally using the Mantoux technique to that of standard Fluzone® administered intramuscularly. The primary objective of the study is to compare the immunogenicity of injected Fluzone® across different dose levels and different routes of administration. The secondary objectives are to describe the number and proportions of subjects in each group experiencing any injection site or systemic symptoms and the proportion of subjects who experience moderate-to-severe symptoms post vaccination. Approximately 31 subjects per group (217 in total) will be enrolled with each group determined by dose and route of administration of vaccines. Subjects will be observed in the clinic for at least 30 minutes after immunization and will maintain a memory aid to record daily oral temperature and any systemic and local reactions for 7 days after the day of immunization. Subjects will be contacted by phone between 8 to 12 days after immunization to review their 7-day memory aid, including the assessment of their recorded daily oral temperature, any local or systemic reactions, and the occurrence of any other AEs and SAEs. Subjects will return at 28 (+/- 3) days after immunization to assess the occurrence of unsolicited AEs and SAEs and complete an acceptability and functional skill questionnaire. Serum for immunogenicity evaluations will be obtained prior to the first vaccination and approximately 28 (+/- 3) days post vaccination. The 2005-2006 formulation will be used for all seven groups.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy, as determined by medical history and clinical assessment before entering the study.
* Between the ages of 18 and 49 (greater than or equal to 18 and less than 50)
* Provides written informed consent
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, menopausal or surgically sterile or negative serum/urine pregnancy test within 24 hours prior to the time of vaccination.

Exclusion Criteria:

* Breast-feeding or pregnant.
* History of receiving 2003-2004, 2004-2005 or 2005-2006 influenza vaccine.
* Known allergy to eggs or other components of the vaccine (e.g., thimerosal).
* History of a severe reaction following influenza vaccination, systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing the same substances.
* History of Guillain-Barre Syndrome.
* Immunosuppression as a result of underlying illness or treatment.
* Use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg per day of beclomethasone dipropionate or equivalent) within 1 month prior to vaccination.
* Use of other immunosuppressive or cytotoxic drugs or radiation therapy within the six months prior to vaccination.
* Active neoplastic disease or history of any hematologic malignancy in the past 5 years (except localized skin or prostate cancer that is stable in the absence of therapy).
* Acute or chronic condition that (in the opinion of the Investigator) would render vaccination unsafe or would interfere with the evaluation of responses including, but not limited to the following: known chronic liver disease, significant renal disease, oxygen-dependent chronic lung disease, New York Heart Association Functional Class III or IV, unstable or progressive neurologic disorder, insulin-treated diabetes mellitus.
* Use of experimental vaccines or medications within the month prior to study entry, or expected use of experimental vaccines or medications during the entire study period after inoculation with study vaccine.
* Use of experimental devices or participation in a medical procedure trial within the month prior to study entry, or expected use of experimental devices or participation in a medical procedure trial during the entire study period.

  13. Receipt of immunoglobulin or other blood product within 3 months prior to enrollment.
* Receipt of other licensed vaccines within the preceding 4 weeks or expected to receive a licensed vaccine within 28 days (prior to visit 2) following trial vaccination.
* Subject is enrolled in a conflicting clinical trial.
* Thrombocytopenia or bleeding disorder or therapy contraindicating IM vaccination.
* Female planning on becoming pregnant within one month of vaccination.
* Acute disease at the time of enrollment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever).
* Febrile illness with temperature greater than or equal to 38 degrees Celsius (100.4 degrees Fahrenheit) within 72 hours prior to enrollment.
* Receipt of allergy shots within the preceding 7 days or expected to receive allergy shots within 7 days following vaccination.
* Any condition that, in the opinion of the investigator, would pose a health risk to the participant.
* Presence of any active skin disease at the injection site that, in the opinion of the Investigator, would impact vaccine delivery or assessment of vaccination site.
* History of drug abuse or alcohol abuse in the five years prior to enrollment.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2005-11; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Immunogenicity evaluated by haemagglutination-inhibition assay (HAI). | Blood sampled at day 28 +/- 3 days post vaccination.

SECONDARY OUTCOMES:
Safety: solicited adverse events (AE)-reactogenicity following each vaccination (local and systemic reactions); unsolicited adverse events, and serious AEs. | Adverse events-reactogenicity following each vaccination. Unsolicited AEs through day 28 +/- 3. Serious AEs occurring during the length of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States